CLINICAL TRIAL: NCT04013373
Title: Home-Based Fluid Status Monitoring in Heart Failure Patients Recently Hospitalized for Acute Heart Failure
Brief Title: Home-Based Fluid Status Monitoring in Heart Failure Patients
Status: Terminated | Type: Observational
Why Stopped: Covid-19 pandemic
Sponsor: ImpediMed Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IPD-HBHF-001
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- BIS home-based monitoring
  Interventions: Device: SOZO Bioimpedance Spectroscopy Device

INTERVENTIONS:
Device: SOZO Bioimpedance Spectroscopy Device — Bioimpedance spectroscopy measurements for assessment of fluid status

SUMMARY:
This is a prospective, multi-center, single-arm study enrolling adult patients who have been hospitalized for heart failure and subsequently discharged. For the duration of study participation, patients will obtain daily at-home bioimpedance measurements. Heart failure symptoms, medications, and re-hospitalizations will be tracked. Additionally, quality of life questionnaires will be administered at the beginning and end of study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or older
2. NYHA Class II or III at the time of study enrollment
3. Undergoing discharge following hospitalization for acute heart failure
4. Planned continued treatment for heart failure
5. Patient is able to stand or sit upright for bioimpedance spectroscopy measurements
6. Patient reports access to reliable Wi-Fi connection at home
7. Patient reports adequate space for the SOZO device at home
8. Patient provides written informed consent and authorization to use and disclose health information, including willingness to comply with study procedures

Exclusion Criteria:

1. Patient has an implanted cardiac rhythm management device (pacemaker or implantable cardioverter defibrillator)
2. Patient has a confirmed diagnosis of acute coronary syndrome during current admission
3. Patient is enrolled in a concurrent interventional study of an experimental treatment that may confound the results of this study, in the investigator's opinion
4. Patient has a clinical condition that would not allow them to complete the study
5. Patient has had surgical revascularization using saphenous vein grafting that may affect venous return
6. Patient is pregnant or lactating
7. Patient has nephrotic syndrome or nephrosis
8. Patient has end-stage renal disease requiring chronic dialysis
9. Patient has been diagnosed with lymphedema
10. Patient has chronic liver failure or cirrhosis
11. Patient has been diagnosed with thrombophlebitis or deep vein thrombosis in arms or legs in the past 90 days
12. Patient has an amputation of a limb [Exception: amputation of digits may not affect bioimpedance spectroscopy measurements and will be permitted at the discretion of the study sponsor]
13. Patient has any other medical condition that, in the opinion of the investigator, will impair the subject's ability to complete study procedures or participate in the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are being discharged home from a hospitalization for heart failure
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Serial bioimpedance spectroscopy (BIS) measurements including extracellular fluid and total body water | 45 days
  Characterize BIS trends that precede hospital readmissions for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: James T Heywood, MD, Principal Investigator — Scripps Clinic
Locations (15):
- United States (15):
  - Alliance Research Institute, Canoga Park, California
  - Du Cardiology, Encinitas, California
  - San Diego Cardiovascular Associates, Encinitas, California
  - SC Clinical Research, Garden Grove, California
  - Scripps Clinic, John R. Anderson V Medical Pavilion, La Jolla, California
  - MD Strategies Research Centers, National City, California
  - Heart Care Associates, Oceanside, California
  - Blue Coast Cardiology, Vista, California
  - Research Alliance, Clearwater, Florida
  - Infinite Clinical Research, Doral, Florida
  - International Research Associates, Miami, Florida
  - Amavita Health, North Miami Beach, Florida
  - Broward Research Center, Pembroke Pines, Florida
  - Flint Cardiovascular, Flint, Michigan
  - Sierra Clinical Research, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Accardi AJ, Matsubara BS, Gaw RL, Daleiden-Burns A, Heywood JT. Clinical Utility of Fluid Volume Assessment in Heart Failure Patients Using Bioimpedance Spectroscopy. Front Cardiovasc Med. 2021 Apr 7;8:636718. doi: 10.3389/fcvm.2021.636718. eCollection 2021. PMID 33898536